CLINICAL TRIAL: NCT07242820
Title: Reducing Neoplasia Recurrence After Non-thermal Endoscopic Resection of Large Colorectal Polyps
Acronym: COSA-RCT
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Centre hospitalier de l'Université de Montréal (CHUM) (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: 2026-13165
Record Dates: First submitted 2025-11-17; First posted 2025-11-21 (Actual); Last update posted 2025-11-21 (Actual); Status verified 2025-11

CONDITIONS: Colorectal Cancer; Polyp of Colon
MeSH Terms: conditions — Colorectal Neoplasms; Colonic Polyps

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Endoscopic mucosal resection (EMR) + adjuvant thermal ablation (Experimental): Adjuvant thermal ablation will be applied to the base and outside margins of the resection site after non-thermal EMR.
  Interventions: Procedure: Adjuvant thermal ablation
- Endoscopic mucosal resection (EMR) (Active Comparator): After non-thermal EMR, no adjuvant thermal ablation will be performed.
  Interventions: Procedure: No adjuvant thermal ablation

INTERVENTIONS:
Procedure: Adjuvant thermal ablation — When the endoscopist determines that the resection is complete, submucosal injection (0.9% NaCl with methylene blue solution) using the h-APC probe (ERBEJET 2 attached to Vio3 electrosurgical unit, pressure: 40 bar) will be performed to further expose the resection margin. Adjuvant thermal ablation will be applied to the outside margins of the resection site using the h-APC probe.
  Adjuvant thermal ablation will then also be applied to the base of the resection site using the h-APC probe. The precise electrocautery mode (PRECISE-APC setting 9) will be used to apply thermal ablation, as previously described for h-APC.
  Arms: Endoscopic mucosal resection (EMR) + adjuvant thermal ablation
Procedure: No adjuvant thermal ablation — After performing non-thermal EMR with thermal ablation, adjuvant thermal ablation will not be performed.
  Arms: Endoscopic mucosal resection (EMR)

SUMMARY:
The goal of this clinical trial is to clarify the role of adjuvant thermal ablation for non-thermal endoscopic mucosal resection (EMR) of large (≥20mm) flat colorectal polyps (so-called laterally spreading lesions [LSLs]).

The hypothesis is that adding adjuvant thermal ablation to non-thermal EMR (vs no ablation) will result in lower lesion recurrence rates at 6-month follow-up, and non-inferior adverse events (AE) rates 14 days post EMR.

For participants with planned EMR, endoscopists will perform non-thermal EMRs as per standard of care and:

* adjuvant thermal ablation will either not be performed (control group), or will be applied to the base and outside margins of the resection site (experimental group);
* then, all patients will be contacted 14-44 days after EMR, to verbally ascertain the occurrence of AEs;
* then, all patients will undergo a first follow-up colonoscopy at 6 months after initial conoloscopy to assess lesion recurrence;
* finally, all patients will undergo a second and final colonoscopy 18 months after EMR.

DETAILED DESCRIPTION:
This trial is an open-label, two-arm, parallel-group, multicenter RCT with co-primary outcomes (superiority for recurrence, non-inferiority for AEs). Patients undergoing non-thermal EMR will be randomized (1:1) to adjuvant thermal ablation (experimental group) or no ablation (control group).

All participating endoscopists will view dedicated teaching videos of the standard thermal ablation technique and key technical details to ensure consistent study procedures. Patients with planned EMR procedures will be invited by a research assistant before the EMR to participate in the study. Patients will be randomized to control or experimental groups in a 1:1 ratio using a central REDCap randomization module after the EMR resection phase is completed and immediately before adjuvant thermal ablation (intervention). This will limit bias by ensuring that the EMR technique is not affected by group allocation. When 2 or more lesions are present in a patient, the largest lesion will be chosen for inclusion in the study and all lesions will be photodocumented for auditing purposes.

No ablation (control group): Non-thermal EMR will be performed as per standard of care with submucosal injection and non-electrocautery resection of all visually visible polyp tissue using a snare. When the endoscopist determines that the resection is complete, no adjuvant thermal ablation of the post-EMR defect will be performed. Defect closure using clips will be performed only if there is concern for injury to the muscle layer or signs of overt perforation. A tattoo will be placed 3 cm distal to the resected lesion to allow for better identification of the resection site for follow-up. If multiple large polyps are found and removed, the largest lesion (study polyp) will be marked with two tattoos 3 cm distally and 3 cm proximally, to clearly identify the study polyp resection site.

Adjuvant thermal ablation (experimental group): Non-thermal EMR will be performed as per standard of care with submucosal injection and non-electrocautery resection of all visually visible polyp tissue using a snare. When the endoscopist determines that the resection is complete, submucosal injection (0.9% NaCl with methylene blue solution) using the h-APC probe (ERBEJET 2 attached to Vio3 electrosurgical unit, pressure: 40 bar) will be performed to further expose the resection margin. Adjuvant thermal ablation will be applied to the outside margins of the resection site using the h-APC probe. Then, adjuvant thermal ablation will also be applied to the base of the resection site using the h-APC probe. The precise electrocautery mode (PRECISE-APC setting 9) will be used to apply thermal ablation, as previously described for h-APC. Defect closure using clips will be performed only if there is concern for injury to the muscle layer or signs of overt perforation. A tattoo will be placed in the same way as described in the control group and, again, if multiple large polyps are found and removed, the largest lesion (study polyp) will be marked with two tattoos 3 cm distally and 3 cm proximally, to clearly identify the study polyp resection site.

At 6 months after initial colonoscopy, patients will undergo a first follow-up colonoscopy, as suggested by current guidelines and from studies showing that most recurrences occurred within the first 6 months. A window of 3 to 13 months will be permitted for the first follow-up. If recurrence is detected, patients will undergo subsequent colonoscopies at shortened intervals, as determined by the treating endoscopist, until no recurrence is detected. If surgery is performed due to difficulty in treating recurrence, patients will undergo a follow-up colonoscopy 6 months after surgery to detect any possible recurrence. All patients will undergo a second and final study colonoscopy 18 months after randomization, which will also mark the end of study follow-up. The second follow-up may be conducted within a window of 14 to 24 months. Subsequent colonoscopies will then be recommended outside the study as per routine care for such a clinical situation.

ELIGIBILITY:
Inclusion Criteria:

* Adult patients
* Undergoing EMR for large (≥20 mm) colorectal LSL
* Providing written and informed consent for study participation

Exclusion Criteria:

* Inflammatory bowel disease
* Non-elective colonoscopy
* Poor general health (American Society of Anesthesiologists classification >III)
* Coagulopathy or thrombocytopenia (international normalized ration ≥1.5 or platelets <50*10^9/L)
* Bulky lesions (granular mixed with ≥10mm module).

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 752 (Estimated)
Dates: Start 2025-12 (Estimated); Primary Completion 2031-05 (Estimated); Study Completion 2032-05 (Estimated)

PRIMARY OUTCOMES:
Lesion recurrence rate | 6 months
  Defined as the number of cases with pathology-confirmed hyperplastic, serrated, or adenomatous histology at the tattooed resection site compatible with the study polyp histology divided by the total number of cases.
Clinically significant adverse event (AE) rate | 14 days
  Defined as the number of cases with delayed bleeding (blood per rectum resulting in emergency room visit, unplanned hospitalization, endoscopic, radiologic, or surgical intervention) and/or delayed perforation (endoscopic or radiologic evidence of significant air or any luminal contents outside the gastrointestinal tract) divided by the total number of cases.

SECONDARY OUTCOMES:
Any delayed bleeding rate | 14 days
  Defined as the number of cases with blood per rectum, regardless of clinical significance, divided by the total number of cases.
Lesion recurrence rate at 18-month follow-up | 18 months
  Defined as the number of cases with pathology-confirmed hyperplastic, serrated, or adenomatous histology at the tattooed resection site compatible with the study polyp histology divided by the total number of cases.

OTHER OUTCOMES:
High-grade dysplasia rate at the 18-month follow-up | 18 months
  Defined as the number of cases with high-grade dysplasia on resection scars divided by the total number of cases.
Rate of CRC during the 18-month follow-up period | From enrollment to the final follow-up colonoscopy at 18 months
  Defined as the number of cases with pathology-confirmed carcinomas divided by the total number of cases.
Colonoscopies to lesion clearance | 18 months
  Defined as the total number of colonoscopies required to achieve lesion clearance, which means no histologic recurrence at the resection scar on follow-up.
EMR procedure time | 1 day
  Defined as the length of time required for the initial EMR.
Rate of delayed bleeding in the proximal colon | 14 days
  Number of cases with clinically significant delayed bleeding in the proximal colon (proximal to the splenic flexure) divided by the total number of cases.
Defect closure time | 1 day
  Time required for defect closure.
Rate of technical success for complete defect closure | 6 months
  Number of cases with technical success for complete defect closure (defined as adequate apposition of the mucosal defect margins without visible submucosal areas >3mm along the closure line) divided by total number of cases.
Costs associated with procedures | From enrollment to the final follow-up colonoscopy at 18 months
  Total costs required to perform non-thermal EMR with adjuvant thermal ablation or without ablation.

CONTACTS AND LOCATIONS:
Locations (1):
- Centre Hospitalier de l'Université de Montréal, Montreal, Quebec, Canada

IPD SHARING:
Plan to Share IPD: Yes
Individual participant data that underlie the results reported in this article, after deidentification (text, tables, figures and appendices).
Supporting Information: Study Protocol, SAP, ICF, CSR, Analytic Code
Time Frame: Beginning 12 months and ending 36 months following article publication.
Access Criteria: Proposals should be directed to daniel.von.renteln.med@ssss.gouv.qc.ca. To gain access, data requestors will need to sign a data access agreement.